CLINICAL TRIAL: NCT07190274
Title: Impact of Frailty on Risk Prediction, Treatment Strategies, and Short-Term Outcomes in Patients With Acute Coronary Syndrome
Brief Title: Prospective Observational Cohort Study on Impact of Frailty on Risk Prediction, Treatment Strategies, and Short-Term Outcomes in Patients With Acute Coronary Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady Gamal Nabih Habib, Principal Investigator, Assiut University
Other Study IDs: frailty in ACS patients
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Frailty; ACS (Acute Coronary Syndrome); MACE; GRACE Score
Keywords: frailty; ACS
MeSH Terms: conditions — Frailty; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
we aim :

* To evaluate how frailty influences acute management decisions (invasive vs conservative strategy) in ACS patients and whether it independently affects short-term outcomes.
* To determine whether adding frailty assessment to existing ACS risk prediction models improves the prediction of 30-day mortality and major adverse cardiovascular events (MACE) in elderly ACS patients.

DETAILED DESCRIPTION:
Frailty is a geriatric syndrome used to define elderly patients with impaired resistance to stressors due to a decline in physiological reserve. Frailty has become increasingly relevant in the field of cardiovascular medicine, not only for the increased aging of the population, but also for the emerging evidence linking CVD and frailty both at the mechanistic level and the epidemiologic level.

The elderly represent an increasing proportion of ACS patients, but they are often excluded from or underrepresented in clinical trials. A thorough assessment of older ACS patients is important, including the evaluation of frailty or comorbidity from the onset of hospitalization and extending to intervention, medications, and type and frequency of MACE. This strategy enables the delivery of a personalized approach for such a vulnerable subgroup.

While established ACS risk models like the GRACE and TIMI scores guide treatment decisions and predict outcomes, they do not account for frailty, an independent, multidimensional predictor of adverse events in the elderly.

Evaluating both the predictive value of frailty and its effect on treatment decisions and outcomes provides comprehensive insight into its clinical relevance in ACS.

ELIGIBILITY:
Inclusion Criteria:

* Elderly: Age ≥65 years .
* STEMI/NSTEMI (ESC/ACC criteria)
* Presentation <24h of symptom onset

Exclusion Criteria:

* Terminal illness (life expectancy <1 month)
* Severe dementia precluding assessment
* Declined consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of patients aged ≥65 years presenting with STEMI or NSTEMI within 24 hours of symptom onset, excluding those with terminal illness, severe dementia, or refusal of consent.
Sampling Method: Non-Probability Sample
Enrollment: 645 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
30-day Major Adverse Cardiovascular Events (MACE) | 30 days after index admission
  Composite outcome including cardiovascular death, non-fatal myocardial infarction, stroke, or urgent revascularization, stratified by frailty status.

SECONDARY OUTCOMES:
All-cause mortality | 30 days after index admission
  Mortality occurring during index hospitalization
Acute Kidney Injury (AKI) | 30 days after index admission
  AKI defined according to KDIGO criteria (increase in serum creatinine ≥0.3 mg/dL within 48 hours or ≥1.5 times baseline within 7 days).

REFERENCES:
- See also: 1. Cepas-Guillén P, Diez-Villanueva P. One-year clinical events according to frailty in older patients with non-ST elevation acute coronary syndrome undergoing coronary angiography: an analysis of the IMPACT-TIMING-GO study. J Geriatr Cardiol. 2025;22(1) — https://pmc.ncbi.nlm.nih.gov/articles/PMC11937830